CLINICAL TRIAL: NCT07279129
Title: A Pilot Feasibility Study to Integrate PrEP Into Emergency Departments Using Decision Support Tools
Brief Title: Decision Support Tool to Integrate PrEP Into Emergency Departments
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: NCR256674
Record Dates: First submitted 2025-11-06; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: HIV
Keywords: PrEP; Emergency departments; Decision support tools; HIV prevention
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ED-PrEP (Active Comparator): In Phase 1 (Pre-DST) PrEP eligible patients who have agreed to PrEP will receive a PrEP prescription facilitated by a PrEP Champion; there will be no structured engagement intervention (i.e., the DST).
  Interventions: Behavioral: PrEP Delivery
- ED-PrEP + DST (Experimental): In Phase 2 (Post-DST) PrEP Champions will integrate the DST into all patient encounters, facilitating the use of the DST as well as the provision of any identified resources.
  Interventions: Behavioral: Decision support tool; Behavioral: PrEP Delivery

INTERVENTIONS:
Behavioral: Decision support tool — Participants enrolled during Phase 2 will engage in all the activities from Phase 1 and will receive the DST intervention. The DST will be designed and programmed to generate results if tablet-based (or to be easily manually scored if paper-based) to display the participant's PrEP knowledge and intention score, self-efficacy score, level of self-perceived risk, as well as generate a list of unmet needs. Upon completion of the DST, the Champion will review these results and discuss them with the participant. Referrals for needed resources will be proactively provided in the ED. After the DST delivery, participants will receive a PrEP prescription and follow-up appointment with a community PrEP provider.
  Arms: ED-PrEP + DST
Behavioral: PrEP Delivery — Participants enrolled during Phase 1 will receive a 14-day prescription of TDF/FTC or FTC/TAF before leaving the ED and an appointment with a community PrEP provider. The Champion will provide brief HIV prevention and PrEP medication counseling including proper dosing, missed doses, review of medication side effects and efficacy, and risk reduction counseling including condom use. Participants will receive a PrEP information brochure. The Champion will also make the initial appointment with the PrEP community provider for within 7 days of the ED visit. Community PrEP providers will be identified using local resources, CDC PrEP locators, and insurance; appointments will be scheduled according to patient preference. All participants will receive a text message reminder two days prior, and a reminder call one day prior.

SUMMARY:
This project will explore the development of a personalized decision support tool to assist with pre-exposure prophylaxis (PrEP) initiation and persistence among patients identified in the emergency department (ED) and urgent care settings as PrEP eligible. First, the investigators will use a sequence of validated implementation science methodologies to develop and validate a decision support tool designed to optimize PrEP persistence by strengthening self-efficacy by addressing the multifaceted medical and social needs of the individual patient. The investigators will then test the preliminary effectiveness of this tool through a pilot stepped wedge implementation trial in two EDs and an urgent care in Baltimore, MD and Washington, DC among 120 PrEP eligible patients to determine PrEP initiation, linkage to care, persistence, and adherence rates.

DETAILED DESCRIPTION:
Despite its promise, rates of pre-exposure prophylaxis (PrEP) uptake in the United States (US) have been modest. Innovative strategies are needed to improve access to PrEP in venues where patients with a high-risk of HIV acquisition may present for care, such as the Emergency Department (ED) or Urgent Care (UC). Recent pilot studies have tested rapid PrEP initiation at the George Washington University (GWU) ED in Washington, DC, and the Johns Hopkins Hospital (JHH) ED in Baltimore, MD, two priority jurisdictions in the US Ending the HIV Epidemic (EHE) initiative, that contribute to 50% of overall new diagnoses in the U.S. These studies found that a significant proportion of patients in the ED are PrEP eligible (96% at JHU - 60% at GWU), yet only 3% of patients who were eligible successfully initiated PrEP following community referral. Barriers to PrEP implementation were multi-faceted, including structural issues (e.g., limited ED provider time to discuss PrEP), patient issues (e.g., competing medical issues, lack of self-perceived HIV risk), and social determinants (e.g., finance, unstable housing, lack of primary care and transportation). PrEP prescribing in the ED/UC (ED-PrEP), while feasible, will also need to consider the higher vulnerabilities and complex competing needs of patients who present for care in these settings, and thus, PrEP prescriptions must be paired with individualized social support to ensure long-term adherence and persistence beyond the initial ED encounter.

This R34 Clinical Trial Planning Grant aims to enhance PrEP uptake among eligible ED/UC patients by piloting a patient-centered Decision Support Tool (DST) for PrEP prescribing. The project seeks to address barriers such as low HIV risk perception and social needs (e.g., insurance, transportation, housing) using the WHO Social Determinants of Health Framework adapted for PrEP. A "Personalized PrEP Pathway" tool will be developed through barrier/facilitator analysis using the Consolidated Framework for Implementation Research (CFIR) and refined via participatory prototyping. The investigators will also identify implementation strategies to optimize ED-PrEP acceptability. Lastly, the investigators will conduct a pilot trial to measure the clinical effectiveness of the DST intervention and implementation outcomes across three clinically distinct venues: the GWU ED in DC, the JHH ED in Baltimore, and the GWU Cedar Hill Urgent Care (CHUC), a high-volume DC UC with limited HIV resources. The GWU and JHH EDs will build upon existing HIV services, whereas inclusion of CHUC will be critical to determining the scalability of the pilot intervention. The ED-PrEP intervention will have three components: 1) Routine screening for PrEP eligibility and HIV testing; 2) PrEP prescribing by ED/UC providers; and 3) Use of a DST to facilitate PrEP initiation and persistence. A multidisciplinary team of experienced HIV clinicians, emergency medicine and implementation science experts seeks to accomplish the following aims:

Aim 1: Develop a patient-centered decision-support tool (DST) to support ED-based PrEP prescribing. The investigators will conduct in-depth interviews (IDI) using CFIR followed by participatory prototyping with PrEP users (n=30) and key stakeholders (n=20) from the two EDs and local communities. IDIs will identify barriers/facilitators to PrEP uptake at the patient and system levels and inform the development of a "Personalized PrEP Pathway" DST that addresses perceived HIV risk and social determinants. Two participatory prototyping workshops, utilizing the nominal group technique, will be conducted to refine the DST to enhance end-user acceptability.

Aim 2: Determine how to optimize the acceptability of an ED-based PrEP intervention using the Normalization Process Theory (NPT) framework across 12 EDs/UCs in the DC-Baltimore region. Local ED providers and PrEP navigators (n=60) will be recruited to review an asynchronous onboarding package for ED- PrEP. They will then be surveyed using a validated NPT tool to seek feedback on how to optimize intervention acceptability and feasibility. The investigators will then refine the tool and develop implementation support resources.

Aim 3: Determine the preliminary effectiveness of ED-PrEP vs ED-PrEP + DST in increasing ED-based PrEP initiation and persistence. The investigators will conduct a phased implementation trial across the three sites among 120 PrEP-eligible ED patients. Phase 1 participants will receive a standard of care PrEP prescription facilitated by a PrEP Champion. In Phase 2, the Champion will also administer the DST and provide the recommended individual and structural supports. The primary outcome will be PrEP persistence at 4 months post-enrollment; secondary outcomes include PrEP initiation, linkage to care, biological and self-reported adherence at 1- and 4-months. Implementation process outcomes will include the number of eligible patients approached and screened, delivery of onsite HIV testing, volume of PrEP prescribing, and DST completion including the number of resources provided and referrals completed.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Self-report being HIV negative (GWU sites) or are found to be HIV rapid test negative (JHH ED)
* Medically stable ED/UC patients (defined as a triage category level 3, 4, 5 using Emergency Severity Index for ED patients only)

Exclusion Criteria:

* Currently taking PEP, PrEP, or present with signs/symptoms of acute HIV infection
* Pregnant
* Currently taking a nephrotoxic medication
* Diagnosed with medical conditions that are contraindicated with use of TDF/FTC or TAF/FTC
* Have a comorbid medical or psychiatric condition that would make PrEP adherence or ongoing follow-up care difficult
* Admission to the hospital
* Are in police custody/prisoner during the ED visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2027-01-15 (Estimated); Primary Completion 2028-04-15 (Estimated); Study Completion 2028-09-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants who self-report taking PrEP in the past 4 months and have any TFV-DP detected in DBS | 4 months
  PrEP persistence defined as self-report of taking PrEP in the past 4 months and having any TFV-DP detected in DBS

SECONDARY OUTCOMES:
Number of participants who fill a PrEP prescription from the ED | 1 week
  PrEP initiation defined as the number of participants who fill a PrEP prescription from the ED confirmed via EMR
Number of participants who attend a PrEP clinic visit | 1 week
  Initial PrEP linkage defined as the number of participants who attend a clinic visit confirmed via self-report or clinic record
Number of participants who self-report PrEP adherence | 4 months
  PrEP adherence defined as the number of participants who report taking PrEP over the last 4-7 days in a 1-week period
Number of participants with biological PrEP adherence (effective short-term use) | 1 month
  Presence of TFV on urine assay at 1 month
Number of participants with biological PrEP adherence (effective long-term use) | 4 months
  Presence of TFV-DP on DBS test at 4 months

OTHER OUTCOMES:
Proportion of eligible patients approached | from baseline screening in the ED to being approached to be in the study in a 14 month period of time
Proportion of eligible patients tested for HIV | from baseline ED screening to study eligibility in a 14 month period of time
Proportion of eligible patients prescribed PrEP | from screening eligible to discharge from the ED in a 14 month period of time
Proportion who completed the DST intervention | Through study completion at 4 months
  Intervention group
Proportion who completed a PrEP follow-up appointment | 7-10 days after study baseline enrollment
Proportion who received one or more follow-up referral/resources after completing the DST | from the time of DST completion to 1 month after ED discharge
Number of providers who prescribed PrEP across sites | from time of study intervention start to completed enrollment at a site in a 14 month period of time
Number of providers who initiated referrals | from time of study start to time of completion of participant enrollment at site in a 14 month period of time
Number of providers who documented DST use in the EMR | from time of study intervention start to completion of participant enrollment at site in a 14 month period of time
Number of CBOs and services engaged | from time of participant referrals to 1 month post referral in a 14 month period of time
Processes (time/resources) related to community linkage to care | from time of participant referral to 1 month post referral

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - George Washington University Emergency Department, Washington D.C., District of Columbia
  - Johns Hopkins Hospital Emergency Department, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
Participant data may contain sensitive information that would not be appropriate to share with external parties. The Study PIs will review requests that they receive and determine whether a de-identified dataset can be shared in a confidential and anonymous manner.